CLINICAL TRIAL: NCT02502149
Title: A Randomized, Open-Label Study to Evaluate the Pharmacokinetics and Safety of Recombinant Factor VIII Fc Fusion Protein (rFVIIIFc; BIIB031) Manufactured at 15K Scale and at Different Vial Strengths in Previously Treated Subjects With Severe Hemophilia A
Brief Title: Pharmacokinetics and Safety of rFVIIIFc Manufactured at 15,000 L (15K) Scale
Acronym: Elevate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioverativ Therapeutics Inc. (Industry)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 997HA309; 2014-003895-21 (EudraCT Number)
Record Dates: First submitted 2015-05-29; First posted 2015-07-20 (Estimated); Results first posted 2018-04-06 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2018-03

CONDITIONS: Severe Hemophilia A
Keywords: rFVIIIFc; Eloctate; Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — factor VIII-Fc fusion protein; Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rFVIIIFc (15K scale) 1000 IU vial (Experimental): Single injection of rFVIIIFc (current 2K scale) followed by 2 single injections of rFVIIIFc (15K scale) 1000 IU vial at PK2 and PK3 timepoints. Participants will be on prophylaxis regimen along with treatment for bleeding episodes for 26 weeks of treatment period using the rFVIIIFc (15K scale) 1000 IU vial.
  Interventions: Biological: rFVIIIFc
- rFVIIIFc (15K scale) 6000 IU vial (Experimental): Single injection of rFVIIIFc (current 2K scale) followed by 2 single injections of rFVIIIFc high strength vial (15K scale) at PK2 and PK3 timepoints. Participants will be on prophylaxis regimen along with treatment for bleeding episodes for 26 weeks of treatment period using the rFVIIIFc (15K scale) 6000 IU vial.
  Interventions: Biological: rFVIIIFc

INTERVENTIONS:
Biological: rFVIIIFc — As per arm description
  Other Names: Eloctate; BIIB031; efmoroctocog alfa; recombinant coagulation factor VIII Fc fusion protein; antihemophilic factor [recombinant]; Fc fusion protein

SUMMARY:
The primary objective of the study is to compare the pharmacokinetic (PK) of recombinant coagulation factor VIII Fc fusion protein (rFVIIIFc) manufactured at the current scale of 2000 L (2K) to the PK of rFVIIIFc manufactured at the 15,000 L (15K) scale in previously treated participants with severe hemophilia A. The secondary objectives are: to characterize the PK of rFVIIIFc manufactured at the 15K scale at the 15K baseline and after 13 weeks of treatment; to characterize the PK of rFVIIIFc manufactured at the 15K scale at 1000 IU/vial and 6000 IU/vial strengths; and to evaluate the safety of rFVIIIFc manufactured at the 15K scale.

DETAILED DESCRIPTION:
PK assessments are in 3 phases: Pharmacokinetic Assessment 1(PK1): PK assessments following single injection of rFVIIIFc manufactured at the 2K scale. Pharmacokinetic Assessment 2 (PK2): PK assessments are made following a single injection of rFVIIIFc manufactured at the 15K scale where participants are randomized to the 1000 IU vial or 6000 IU/vial strengths. Pharmacokinetic Assessment 3 (PK3): PK assessments are made following 13 weeks of rFVIIIFc treatment manufactured at the 15K scale where participants are randomized to the 1000 IU vial or 6000 IU/vial strengths. After study completion, in countries where rFVIIIFc is not commercially available, eligible participants will be offered enrollment into a long-term safety and efficacy extension study (8HA01EXT [NCT01454739]).

ELIGIBILITY:
Key Inclusion Criteria:

* Have severe hemophilia A, defined as <1 IU/dL (<1%) endogenous FVIII as determined by one-stage clotting assay from the central laboratory at Screening.
* Previously treated subject, defined as having at least 150 documented prior exposure days (EDs) to any recombinant and/or plasma-derived FVIII and/or cryoprecipitate products at Day 1. Fresh frozen plasma treatment must not be considered in the count for documented exposure days.
* No history of a positive inhibitor test or clinical signs of decreased response to FVIII administrations. Family history of inhibitors will not exclude the subject.
* No measurable inhibitor activity using the Nijmegen-modified Bethesda assay (>=0.6 Bethesda Unit per milliliter [BU/mL] is considered positive) at Screening.

Key Exclusion Criteria:

* Current enrollment in any interventional clinical study in which an investigational drug or approved therapy for investigational use is administered within 30 days prior to the Baseline Visit OR prior participation in any of the following Biogen studies: 998HA101 (NCT01027377), 997HA301 (NCT01181128), 8HA02PED (NCT01458106), 997HA307 (NCT02083965), and 8HA01EXT (NCT01454739).
* Previous participation in this study.
* Any concurrent clinically significant major disease that, in the opinion of the Investigator or Biogen, makes the subject unsuitable for participation in the study.
* Other coagulation disorder(s) in addition to hemophilia A.
* History of hypersensitivity or anaphylaxis associated with FVIII or intravenous (IV) immunoglobulin administration.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-08; Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Bioverativ Therapeutics Inc.
Locations (15):
- United States (8):
  - Research Site, Los Angeles, California
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, East Lansing, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Salt Lake City, Utah
  - Research Site, Seattle, Washington
- Australia (3):
  - Research Site, Camperdown, New South Wales
  - Research Site, Melbourne, Victoria
  - Research Site, Murdoch, Western Australia
- New Zealand (4):
  - Research Site, Grafton, Auckland
  - Research Site, Newtown, Wellington Region
  - Research Site, Christchurch
  - Research Site, Hamilton

RESULTS

PARTICIPANT FLOW:
Groups:
- 2K rFVIIIFc (1000 IU/Vial Strength) (PK1): All participants received recombinant factor VIII Fc fusion protein (rFVIIIFc) (1000 IU/vial strength), 50 International Unit per kilogram (IU/kg), manufactured in 2K (2000 liter bioreactor scale) for pharmacokinetic assessment 1 (PK1).
- 15K rFVIIIFc (1000 IU/Vial Strength) (PK2): Participants who received 2K rFVIIIFc 1000 IU/vial (50 IU/kg) for PK1 were randomized to receive rFVIIIFc (1000 IU/vial strength), 50 IU/kg, manufactured in 15K (15000 liter bioreactor scale) for pharmacokinetic assessment 2 (PK2). Following PK2 assessments, participants received prophylactic treatment with any of 5 available 15K vial strengths during the treatment phase. After 13 weeks of treatment with15K rFVIIIFc, participants will be re-evaluated at Pharmacokinetic assessment 3 (PK3) at the same vial strength as in PK2. A minimum of 120 hours of washout was observed prior to the PK2 assessment. Following the PK3 assessment, participants will resume to treatment in the Treatment Period until they complete a total of at least 26 weeks of treatment.
- 15K rFVIIIFc (6000 IU/Vial Strength) (PK2): Participants who received 2K rFVIIIFc 1000 IU/vial (50 IU/kg) for PK1 were randomized to receive rFVIIIFc (6000 IU/vial strength), 50 IU/kg, manufactured in 15K (15000 liter bioreactor scale) for PK2. Following PK2 assessments, participants received prophylactic treatment with any of 5 available 15K vial strengths during the treatment phase. After 13 weeks of treatment with15K rFVIIIFc, participants will be re-evaluated at PK3 at the same vial strength as in PK2. A minimum of 120 hours of washout was observed prior to the PK2 assessment. Following the PK3 assessment, participants will resume to treatment in the Treatment Period until they complete a total of at least 26 weeks of treatment.
- 15K rFVIIIFc (1000 IU/Vial Strength) (PK3): Participants who were randomized to receive 15K rFVIIIFc 1000 IU/vial for PK2 assessment were re-evaluated after 13 weeks on treatment for PK3 assessment at same vial strength.
- 15K rFVIIIFc (6000 IU/Vial Strength) (PK3): Participants who were randomized to receive 15K rFVIIIFc 6000 IU/vial for PK2 assessment were re-evaluated after 13 weeks on treatment for PK3 assessment at same vial strength.
Period: PK1 Assessment Period
Arm/Group | 2K rFVIIIFc (1000 IU/Vial Strength) (PK1) | 15K rFVIIIFc (1000 IU/Vial Strength) (PK2) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK2) | 15K rFVIIIFc (1000 IU/Vial Strength) (PK3) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK3)
Started | 24 | 0 | 0 | 0 | 0
Completed | 24 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Intermediate
Arm/Group | 2K rFVIIIFc (1000 IU/Vial Strength) (PK1) | 15K rFVIIIFc (1000 IU/Vial Strength) (PK2) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK2) | 15K rFVIIIFc (1000 IU/Vial Strength) (PK3) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK3)
Started | 24 | 0 | 0 | 0 | 0
Completed | 23 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Discontinued prematurely | 1 | 0 | 0 | 0 | 0
Period: PK2 Assessment Period
Arm/Group | 2K rFVIIIFc (1000 IU/Vial Strength) (PK1) | 15K rFVIIIFc (1000 IU/Vial Strength) (PK2) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK2) | 15K rFVIIIFc (1000 IU/Vial Strength) (PK3) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK3)
Started | 0 | 11 | 12 | 0 | 0
Completed | 0 | 11 | 12 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Treatment Period
Arm/Group | 2K rFVIIIFc (1000 IU/Vial Strength) (PK1) | 15K rFVIIIFc (1000 IU/Vial Strength) (PK2) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK2) | 15K rFVIIIFc (1000 IU/Vial Strength) (PK3) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK3)
Started | 0 | 0 | 0 | 11 | 12
Completed | 0 | 0 | 0 | 11 | 12
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 2K/15K rFVIIIFc (1000/6000 IU/Vial Strength)- All Participants: All participants received rFVIIIFc (1000 IU/vial strength), 50 IU/kg, manufactured in 2K (2000 liter bioreactor scale) for PK1. At PK1, participants were randomized to receive rFVIIIFc (1000 or 6000 IU/vial strength), 50 IU/kg, manufactured in 15K (15000 liter bioreactor scale) for PK2. Following PK2 assessments, participants received prophylactic treatment with any of 5 available 15K vial strengths during the treatment phase. After 13 weeks of treatment with 15K rFVIIIFc, participants were re-evaluated at PK3 at the same vial strength as in PK2. A minimum of 120 hours of washout was observed prior to the PK2 assessment. Following the PK3 assessment, participants will resume to treatment in the Treatment Period until they complete a total of at least 26 weeks of treatment.
Arm/Group | 2K/15K rFVIIIFc (1000/6000 IU/Vial Strength)- All Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (12.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Not reported | 17

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf) as Measured by One-stage Activated Partial Thromboplastin Time (aPTT) Clotting Assay for Pharmacokinetic Assessment 1 (PK1) and Pharmacokinetic Assessment 2 (PK2)
Description: AUCinf is area under the concentration-time curve from time zero to infinity. Results were summarized overall for 15K rFVIIIFc 1000 IU/vial and 6000 IU/Vial (PK2).
Time Frame: Pre-dose and post dose at: 0.5 hour (hr), 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The Pharmacokinetic Analysis Set (PKAS) included all participants who have evaluable PK profiles. All 24 participants had data available from PK1 and/or PK2 and were included in the analysis model for this outcome. Hence, the data for 24 participants has been reported for PK2.
Measure: Geometric Mean (90% Confidence Interval); unit: International unit*hour per deciliter
Groups:
- 2K rFVIIIFc (1000 IU/Vial Strength) (PK1): All participants received rFVIIIFc (1000 IU/vial strength), 50 IU/kg, manufactured in 2K (2000 liter bioreactor scale) for pharmacokinetic assessment 1 (PK1).
  .
- 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2): Participants who received 2K rFVIIIFc 1000 IU/vial (50 IU/kg) for PK1 were randomized to receive rFVIIIFc (1000 or 6000 IU/vial strength), 50 IU/kg, manufactured in 15K (15000 liter bioreactor scale) for pharmacokinetic assessment 2 (PK2). Following PK2 assessments, participants received prophylactic treatment with any of 5 available 15K vial strengths during the treatment phase. After 13 weeks of treatment with 15K rFVIIIFc, participants were re-evaluated at Pharmacokinetic assessment 3 (PK3) at the same vial strength as in PK2. A minimum of 120 hours of washout was observed prior to the PK2 assessment. Following the PK3 assessment, participants were resumed to treatment in the Treatment Period until they complete a total of at least 26 weeks of treatment.
Arm/Group | 2K rFVIIIFc (1000 IU/Vial Strength) (PK1) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2)
Number analyzed (Participants) | 24 | 24
International unit*hour per deciliter | 2255.6 [1886.2 to 2697.4] | 2425.8 [2084.2 to 2823.4]
Statistical Analysis 1: Comparison: 2K rFVIIIFc (1000 IU/Vial Strength) (PK1) vs 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2); Test type: Other; Adjusted Geometric Mean Ratio = 1.08, 90% CI 2-sided [0.93 to 1.24] — The adjusted geometric mean ratio is calculated as 15K (PK2)/2K (PK1)

2. Primary Outcome: Incremental Recovery (IR) as Measured by One-stage aPTT Clotting Assay for PK1 and PK2
Description: Incremental Recovery is defined as the increase in the circulating FVIII activity in international unit per deciliter (IU/dL) per unit dose administered in international unit per kilogram (IU/kg) (IU/dL per IU/kg). Results were summarized overall for 15K rFVIIIFc 1000 IU/vial and 6000 IU/Vial (PK2).
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS included all participants who have evaluable PK profiles. All 24 participants had data available from PK1 and/or PK2 and were included in the analysis model for this outcome. Hence, the data for 24 participants has been reported for PK2.
Measure: Geometric Mean (90% Confidence Interval); unit: IU/dL per IU/kg
Groups:
- 2K rFVIIIFc (1000 IU/Vial Strength) (PK1): All participants received rFVIIIFc (1000 IU/vial strength), 50 IU/kg, manufactured in 2K (2000 liter bioreactor scale) for pharmacokinetic assessment 1 (PK1).
- 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2): Participants who received 2K rFVIIIFc 1000 IU/vial (50 IU/kg) for PK1 were randomized to receive rFVIIIFc (1000 or 6000 IU/vial strength), 50 IU/kg, manufactured in 15K (15000 liter bioreactor scale) for PK2. Following PK2 assessments, participants received prophylactic treatment with any of 5 available 15K vial strengths during the treatment phase. After 13 weeks of treatment with 15K rFVIIIFc, participants were re-evaluated at PK3 at the same vial strength as in PK2. A minimum of 120 hours of washout was observed prior to the PK2 assessment. Following the PK3 assessment, participants were resumed to treatment in the Treatment Period until they complete a total of at least 26 weeks of treatment.
Arm/Group | 2K rFVIIIFc (1000 IU/Vial Strength) (PK1) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2)
Number analyzed (Participants) | 24 | 24
IU/dL per IU/kg | 2.684 [2.364 to 3.049] | 2.700 [2.458 to 2.964]
Statistical Analysis 1: Comparison: 2K rFVIIIFc (1000 IU/Vial Strength) (PK1) vs 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2); Test type: Other; Adjusted Geometric Mean Ratio = 1.01, 90% CI 2-sided [0.87 to 1.16] — The adjusted geometric mean ratio is calculated as 15K (PK2)/2K (PK1)

3. Secondary Outcome: Maximum Activity (Cmax) of rFVIIIFc as Measured by One-stage aPTT Clotting Assay for PK1 and PK2
Description: Cmax is defined as maximum activity of rFVIIIFc. Results were summarized overall for 15K rFVIIIFc 1000 IU/vial and 6000 IU/Vial (PK2).
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles. All 24 participants had data available from PK1 and/or PK2 and were included in the analysis model for this outcome. Hence, the data for 24 participants has been reported for PK2.
Measure: Geometric Mean (95% Confidence Interval); unit: International units per deciliter (IU/dL
Arm/Group | 2K rFVIIIFc (1000 IU/Vial Strength) (PK1) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2)
Number analyzed (Participants) | 24 | 24
International units per deciliter (IU/dL | 133.20 [123.00 to 144.24] | 134.67 [121.46 to 149.32]

4. Secondary Outcome: Half-life (t½) of rFVIIIFc as Measured by One-stage aPTT Clotting Assay for PK1 and PK2
Description: Half-life is time required for the concentration of the drug to reach half of its original value. Results were summarized overall for 15K 1000 IU/vial and 6000 IU/Vial (PK2).
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Hours (h)
Arm/Group | 2K rFVIIIFc (1000 IU/Vial Strength) (PK1) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2)
Number analyzed (Participants) | 24 | 24
Hours (h) | 14.229 [12.458 to 16.252] | 14.771 [12.910 to 16.900]

5. Secondary Outcome: Clearance (CL) of rFVIIIFc as Measured by One-stage aPTT Clotting Assay for PK1 and PK2
Description: Clearance (CL) is a quantitative measure of the rate at which a drug substance is removed from the body.The total systemic clearance after intravenous dose was estimated by dividing the total administered dose by the plasma Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]). Results were summarized overall for 15K rFVIIIFc 1000 IU/vial and 6000 IU/Vial (PK2).
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: milliliter per hour per kilogram(mL/h/kg
Arm/Group | 2K rFVIIIFc (1000 IU/Vial Strength) (PK1) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2)
Number analyzed (Participants) | 24 | 24
milliliter per hour per kilogram(mL/h/kg | 2.1847 [1.8943 to 2.5198] | 2.0420 [1.7421 to 2.3935]

6. Secondary Outcome: Volume of Distribution at Steady State (Vss) of rFVIIIFc as Measured by One-stage aPTT Clotting Assay for PK1 and PK2
Description: Vss is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state which is estimated by (D/AUC[0-infinity])*(AUMC[0-infinity])/AUC[0-infinity]) where D is the dose of study drug, AUMC(0-infinity) is the area under the first moment curve extrapolated to infinity and AUC(0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time. Results were summarized overall for 15K rFVIIIFc 1000 IU/vial and 6000 IU/Vial (PK2).
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: milliliter per kilogram (mL/kg)
Arm/Group | 2K rFVIIIFc (1000 IU/Vial Strength) (PK1) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2)
Number analyzed (Participants) | 24 | 24
milliliter per kilogram (mL/kg) | 43.80 [40.70 to 47.14] | 43.01 [39.69 to 46.61]

7. Secondary Outcome: Mean Residence Time (MRT) of rFVIIIFc as Measured by One-stage aPTT Clotting Assay for PK1 and PK2
Description: The Mean Residence Time (MRT) is the average time at which the number of absorbed molecules reside in the body, after single-dose administration, and calculated as area under the first moment curve AUMC (0-infinity)/Area Under the Plasma Concentration-Time Curve AUC (0-infinity), where AUMC (0-infinity) is area under the plasma concentration-time first moment curve from time zero to infinite time and AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time. Results were summarized overall for 15K rFVIIIFc 1000 IU/vial and 6000 IU/Vial (PK2).
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: hours (h)
Arm/Group | 2K rFVIIIFc (1000 IU/Vial Strength) (PK1) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2)
Number analyzed (Participants) | 24 | 24
hours (h) | 20.048 [17.561 to 22.887] | 21.063 [18.501 to 23.980]

8. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf) as Measured by One-stage aPTT Clotting Assay for PK2 and PK3
Description: AUCinf is area under the concentration-time curve from time zero to infinity. Results were summarized overall for 15K rFVIIIFc 1000 IU/Vial and 6000 IU/Vial for PK2 and PK3.
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL
Groups:
- 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK3): Participants who were randomized to receive 15K rFVIIIFc 1000 or 6000 IU/vial for PK2 assessment were re-evaluated after 13 weeks on treatment for PK3 assessment at same vial strength.
Arm/Group | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK3)
Number analyzed (Participants) | 23 | 21
IU*h/dL | 2448.6 [2089.0 to 2870.1] | 2697.8 [2295.1 to 3171.0]

9. Secondary Outcome: Incremental Recovery (IR) as Measured by One-stage aPTT Clotting Assay for PK2 and PK3
Description: Incremental Recovery is defined as the increase in the circulating FVIII activity in IU/dL per unit dose administered in IU/kg (IU/dL per IU/kg). Results were summarized overall for 15K rFVIIIFc 1000 IU/Vial and 6000 IU/Vial for PK2 and PK3.
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL per IU/kg
Arm/Group | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK3)
Number analyzed (Participants) | 23 | 23
IU/dL per IU/kg | 2.693 [2.429 to 2.986] | 2.804 [2.588 to 3.038]

10. Secondary Outcome: Maximum Activity (Cmax) of rFVIIIFc as Measured by One-stage aPTT Clotting Assay for PK2 and PK3
Description: Cmax is defined as maximum activity of rFVIIIFc. Results were summarized overall for 15K rFVIIIFc 1000 IU/Vial and 6000 IU/Vial for PK2 and PK3.
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL
Arm/Group | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK3)
Number analyzed (Participants) | 23 | 23
IU/dL | 134.67 [121.46 to 149.32] | 140.38 [129.62 to 152.04]

11. Secondary Outcome: Half-life (t½) of rFVIIIFc as Measured by One-stage aPTT Clotting Assay for PK2 and PK3
Description: Time required for the concentration of the drug to reach half of its original value. Results were summarized overall for 15K rFVIIIFc 1000 IU/Vial and 6000 IU/Vial for PK2 and PK3.
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Hours (h)
Arm/Group | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK3)
Number analyzed (Participants) | 23 | 21
Hours (h) | 14.771 [12.910 to 16.900] | 15.493 [13.625 to 17.617]

12. Secondary Outcome: Clearance (CL) of rFVIIIFc as Measured by One-stage aPTT Clotting Assay for PK2 and PK3
Description: Clearance (CL) is a quantitative measure of the rate at which a drug substance is removed from the body.The total systemic clearance after intravenous dose was estimated by dividing the total administered dose by the plasma Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]). Results were summarized overall for 15K rFVIIIFc 1000 IU/Vial and 6000 IU/Vial for PK2 and PK3.
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: mL/h/kg
Arm/Group | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK3)
Number analyzed (Participants) | 23 | 21
mL/h/kg | 2.0420 [1.7421 to 2.3935] | 1.8556 [1.5786 to 2.1813]

13. Secondary Outcome: Volume of Distribution at Steady State (Vss) of rFVIIIFc as Measured by One-stage aPTT Clotting Assay for PK2 and PK3
Description: Vss is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state which is estimated by (D/AUC[0-infinity])*(AUMC[0-infinity])/AUC[0-infinity]) where D is the dose of study drug, AUMC(0-infinity) is the area under the first moment curve extrapolated to infinity and AUC(0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time. Results were summarized overall for 15K rFVIIIFc 1000 IU/Vial and 6000 IU/Vial for PK2 and PK3.
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg
Arm/Group | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK3)
Number analyzed (Participants) | 23 | 21
mL/kg | 43.01 [39.69 to 46.61] | 40.19 [37.44 to 43.14]

14. Secondary Outcome: Mean Residence Time (MRT) of rFVIIIFc as Measured by One-stage aPTT Clotting Assay for PK2 and PK3
Description: The Mean Residence Time (MRT) is the average time at which the number of absorbed molecules reside in the body, after single-dose administration, and calculated as area under the first moment curve AUMC (0-infinity)/Area Under the Plasma Concentration-Time Curve AUC (0-infinity), where AUMC (0-infinity) is area under the plasma concentration-time first moment curve from time zero to infinite time and AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time. Results were summarized overall for 15K rFVIIIFc 1000 IU/Vial and 6000 IU/Vial for PK2 and PK3.
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: hours (h)
Arm/Group | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK3)
Number analyzed (Participants) | 23 | 21
hours (h) | 21.063 [18.501 to 23.980] | 21.657 [18.877 to 24.847]

15. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf) as Measured by One-stage aPTT Clotting Assay for PK2 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: AUCinf is area under the concentration-time curve from time zero to infinity.
Time Frame: Pre-dose and post dose at: 0.5 hour (hr), 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL
Groups:
- 15K rFVIIIFc (1000 IU/Vial Strength) (PK2): Participants who received 2K rFVIIIFc 1000 IU/vial (50 IU/kg) for PK1 were randomized to receive rFVIIIFc (1000 IU/vial strength), 50 IU/kg, manufactured in 15K (15000 liter bioreactor scale) for PK2. Following PK2 assessments, participants received prophylactic treatment with any of 5 available 15K vial strengths during the treatment phase. After 13 weeks of treatment with 15K rFVIIIFc, participants were re-evaluated at PK3 at the same vial strength as in PK2. A minimum of 120 hours of washout was observed prior to the PK2 assessment. Following the PK3 assessment, participants were resumed to treatment in the Treatment Period until they complete a total of at least 26 weeks of treatment.
- 15K rFVIIIFc (6000 IU/Vial Strength) (PK2): Participants who received 2K rFVIIIFc 1000 IU/vial (50 IU/kg) for PK1 were randomized to receive rFVIIIFc (6000 IU/vial strength), 50 IU/kg, manufactured in 15K (15000 liter bioreactor scale) for PK2. Following PK2 assessments, participants received prophylactic treatment with any of 5 available 15K vial strengths during the treatment phase. After 13 weeks of treatment with 15K rFVIIIFc, participants were re-evaluated at PK3 at the same vial strength as in PK2. A minimum of 120 hours of washout was observed prior to the PK2 assessment. Following the PK3 assessment, participants were resumed to treatment in the Treatment Period until they complete a total of at least 26 weeks of treatment.
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK2) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK2)
Number analyzed (Participants) | 11 | 12
IU*h/dL | 2356.8 [1950.4 to 2847.9] | 2535.8 [1915.6 to 3356.8]

16. Secondary Outcome: Incremental Recovery (IR) of rFVIIIFc as Measured by One-stage aPTT Clotting Assay for PK2 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: Incremental Recovery is defined as the increase in the circulating FVIII activity in international unit per deciliter (IU/dL) per unit dose administered in international unit per kilogram (IU/kg) (IU/dL per IU/kg).
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL per IU/kg
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK2) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK2)
Number analyzed (Participants) | 11 | 12
IU/dL per IU/kg | 2.614 [2.186 to 3.126] | 2.768 [2.408 to 3.181]

17. Secondary Outcome: Maximum Activity (Cmax) of rFVIIIFc as Measured by One-stage aPTT Clotting Assay for PK2 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: Cmax is defined as maximum activity of rFVIIIFc.
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK2) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK2)
Number analyzed (Participants) | 11 | 12
IU/dL | 130.73 [109.33 to 156.31] | 138.40 [120.42 to 159.06]

18. Secondary Outcome: Half-life (t½) of rFVIIIFc as Measured by One-stage aPTT Clotting Assay for PK2 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: Time required for the concentration of the drug to reach half of its original value.
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: Hours (h)
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK2) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK2)
Number analyzed (Participants) | 11 | 12
Hours (h) | 14.118 [11.469 to 17.379] | 15.395 [12.555 to 18.879]

19. Secondary Outcome: Clearance (CL) of rFVIIIFc as Measured by One-stage aPTT Clotting Assay for PK2 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: Clearance (CL) is a quantitative measure of the rate at which a drug substance is removed from the body.The total systemic clearance after intravenous dose was estimated by dividing the total administered dose by the plasma Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]).
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: mL/h/kg
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK2) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK2)
Number analyzed (Participants) | 11 | 12
mL/h/kg | 2.1215 [1.7557 to 2.5635] | 1.9718 [1.4895 to 2.6101]

20. Secondary Outcome: Volume of Distribution at Steady State (Vss) of rFVIIIFc as Measured by One-stage aPTT Clotting Assay for PK2 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: Vss is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state which is estimated by (D/AUC[0-infinity])*(AUMC[0-infinity])/AUC[0-infinity]) where D is the dose of study drug, AUMC(0-infinity) is the area under the first moment curve extrapolated to infinity and AUC(0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time.
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK2) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK2)
Number analyzed (Participants) | 11 | 12
mL/kg | 42.61 [37.28 to 48.71] | 43.38 [38.66 to 48.67]

21. Secondary Outcome: Mean Residence Time (MRT) of rFVIIIFc as Measured by One-stage aPTT Clotting Assay for PK2 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: The Mean Residence Time (MRT) is the average time at which the number of absorbed molecules reside in the body, after single-dose administration, and calculated as area under the first moment curve AUMC (0-infinity)/Area Under the Plasma Concentration-Time Curve AUC (0-infinity), where AUMC (0-infinity) is area under the plasma concentration-time first moment curve from time zero to infinite time and AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time.
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: hours (h)
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK2) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK2)
Number analyzed (Participants) | 11 | 12
hours (h) | 20.087 [16.333 to 24.704] | 22.000 [18.193 to 26.603]

22. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf) as Measured by One-stage aPTT Clotting Assay for PK3 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: AUCinf is area under the concentration-time curve from time zero to infinity.
Time Frame: Pre-dose and post dose at: 0.5 hour (hr), 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK3) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK3)
Number analyzed (Participants) | 9 | 12
IU*h/dL | 2634.5 [2079.8 to 3337.1] | 2746.3 [2130.5 to 3539.9]

23. Secondary Outcome: Incremental Recovery (IR) of rFVIIIFc as Measured by One-stage aPTT Clotting Assay for PK3 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: as for outcome 16
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL per IU/kg
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK3) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK3)
Number analyzed (Participants) | 11 | 12
IU/dL per IU/kg | 2.623 [2.343 to 2.936] | 2.982 [2.650 to 3.355]

24. Secondary Outcome: Maximum Activity (Cmax) of rFVIIIFc as Measured by One-stage aPTT Clotting Assay for PK3 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: Cmax is defined as maximum activity of rFVIIIFc.
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK3) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK3)
Number analyzed (Participants) | 11 | 12
IU/dL | 131.15 [117.18 to 146.80] | 149.41 [132.99 to 167.86]

25. Secondary Outcome: Half-life (t½) of rFVIIIFc as Measured by One-stage aPTT Clotting Assay for PK3 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: Time required for the concentration of the drug to reach half of its original value.
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Hours (h)
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK3) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK3)
Number analyzed (Participants) | 9 | 12
Hours (h) | 15.599 [12.925 to 18.826] | 15.414 [12.593 to 18.868]

26. Secondary Outcome: Clearance (CL) of rFVIIIFc as Measured by One-stage aPTT Clotting Assay for PK3 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: as for outcome 19
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: mL/h/kg
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK3) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK3)
Number analyzed (Participants) | 9 | 12
mL/h/kg | 1.8979 [1.4983 to 2.4041] | 1.8246 [1.4151 to 2.3524]

27. Secondary Outcome: Volume of Distribution at Steady State (Vss) of rFVIIIFc as Measured by One-stage aPTT Clotting Assay for PK3 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: as for outcome 20
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK3) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK3)
Number analyzed (Participants) | 9 | 12
mL/kg | 42.12 [36.95 to 48.02] | 38.80 [35.47 to 42.43]

28. Secondary Outcome: Mean Residence Time (MRT) of rFVIIIFc as Measured by One-stage aPTT Clotting Assay for PK3 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: as for outcome 21
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: hours (h)
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK3) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK3)
Number analyzed (Participants) | 9 | 12
hours (h) | 22.193 [17.923 to 27.480] | 21.264 [17.247 to 26.216]

29. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf) as Measured by the Two-stage Chromogenic Assay for PK1 and PK2
Description: as for outcome 1
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL
Arm/Group | 2K rFVIIIFc (1000 IU/Vial Strength) (PK1) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2)
Number analyzed (Participants) | 24 | 24
IU*h/dL | 2386.4 [2124.1 to 2681.0] | 2777.6 [2453.0 to 3145.2]

30. Secondary Outcome: Incremental Recovery (IR) as Measured by the Two-stage Chromogenic Assay for PK1 and PK2
Description: Incremental Recovery is defined as the increase in the circulating FVIII activity in IU/dL per unit dose administered in IU/kg (IU/dL per IU/kg). Results were summarized overall for 15K rFVIIIFc 1000 IU/vial and 6000 IU/Vial (PK2).
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL per IU/kg
Arm/Group | 2K rFVIIIFc (1000 IU/Vial Strength) (PK1) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2)
Number analyzed (Participants) | 24 | 24
IU/dL per IU/kg | 2.807 [2.412 to 3.267] | 3.253 [2.910 to 3.636]

31. Secondary Outcome: Maximum Activity (Cmax) of rFVIIIFc as Measured by the Two-stage Chromogenic Assay for PK1 and PK2
Description: as for outcome 3
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL
Arm/Group | 2K rFVIIIFc (1000 IU/Vial Strength) (PK1) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2)
Number analyzed (Participants) | 24 | 24
IU/dL | 140.36 [120.61 to 163.34] | 162.73 [145.61 to 181.86]

32. Secondary Outcome: Half-life (t½) of rFVIIIFc as Measured by the Two-stage Chromogenic Assay for PK1 and PK2
Description: Time required for the concentration of the drug to reach half of its original value. Results were summarized overall for 15K rFVIIIFc 1000 IU/vial and 6000 IU/Vial (PK2).
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Hours (h)
Arm/Group | 2K rFVIIIFc (1000 IU/Vial Strength) (PK1) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2)
Number analyzed (Participants) | 24 | 24
Hours (h) | 17.312 [15.840 to 18.921] | 18.146 [15.980 to 20.605]

33. Secondary Outcome: Clearance (CL) of rFVIIIFc as Measured by the Two-stage Chromogenic Assay for PK1 and PK2
Description: as for outcome 5
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: mL/h/kg
Arm/Group | 2K rFVIIIFc (1000 IU/Vial Strength) (PK1) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2)
Number analyzed (Participants) | 24 | 24
mL/h/kg | 2.0952 [1.8649 to 2.3539] | 1.8001 [1.5897 to 2.0383]

34. Secondary Outcome: Volume of Distribution at Steady State (Vss) of rFVIIIFc as Measured by the Two-stage Chromogenic Assay for PK1 and PK2
Description: as for outcome 6
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg
Arm/Group | 2K rFVIIIFc (1000 IU/Vial Strength) (PK1) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2)
Number analyzed (Participants) | 24 | 24
mL/kg | 46.87 [41.48 to 52.96] | 42.02 [37.96 to 46.51]

35. Secondary Outcome: Mean Residence Time (MRT) of rFVIIIFc as Measured by the Two-stage Chromogenic Assay for PK1 and PK2
Description: as for outcome 7
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: hours (h)
Arm/Group | 2K rFVIIIFc (1000 IU/Vial Strength) (PK1) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2)
Number analyzed (Participants) | 24 | 24
hours (h) | 22.370 [19.921 to 25.120] | 23.342 [20.472 to 26.615]

36. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf) as Measured by the Two-stage Chromogenic Assay for PK2 and PK3
Description: as for outcome 8
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL
Arm/Group | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK3)
Number analyzed (Participants) | 23 | 20
IU*h/dL | 2777.6 [2453.0 to 3145.2] | 2754.9 [2312.2 to 3282.4]

37. Secondary Outcome: Incremental Recovery (IR) as Measured by the Two-stage Chromogenic Assay for PK2 and PK3
Description: as for outcome 9
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL per IU/kg
Arm/Group | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK3)
Number analyzed (Participants) | 23 | 23
IU/dL per IU/kg | 3.253 [2.910 to 3.636] | 2.956 [2.656 to 3.289]

38. Secondary Outcome: Maximum Activity (Cmax) of rFVIIIFc as Measured by the Two-stage Chromogenic Assay for PK2 and PK3
Description: as for outcome 10
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL
Arm/Group | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK3)
Number analyzed (Participants) | 23 | 23
IU/dL | 162.73 [145.61 to 181.86] | 147.97 [133.02 to 164.60]

39. Secondary Outcome: Half-life (t½) of rFVIIIFc as Measured by the Two-stage Chromogenic Assay for PK2 and PK3
Description: as for outcome 11
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Hours (h)
Groups:
- 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK3): Participants who were randomized to receive 15K rFVIIIFc 1000 and 6000 IU/vial for PK2 assessment were re-evaluated after 13 weeks on treatment for PK3 assessment at same vial strength.
Arm/Group | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK3)
Number analyzed (Participants) | 23 | 20
Hours (h) | 18.146 [15.980 to 20.605] | 17.289 [15.078 to 19.823]

40. Secondary Outcome: Clearance (CL) of rFVIIIFc as Measured by the Two-stage Chromogenic Assay for PK2 and PK3
Description: as for outcome 12
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: mL/h/kg
Arm/Group | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK3)
Number analyzed (Participants) | 23 | 20
mL/h/kg | 1.8001 [1.5897 to 2.0383] | 1.8173 [1.5251 to 2.1654]

41. Secondary Outcome: Volume of Distribution at Steady State (Vss) of rFVIIIFc as Measured the Two-stage Chromogenic Assay for PK2 and PK3
Description: as for outcome 13
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg
Arm/Group | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK3)
Number analyzed (Participants) | 23 | 20
mL/kg | 42.02 [37.96 to 46.51] | 40.59 [36.01 to 45.75]

42. Secondary Outcome: Mean Residence Time (MRT) of rFVIIIFc as Measured by the Two-stage Chromogenic Assay for PK2 and PK3
Description: as for outcome 14
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: hours (h)
Arm/Group | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK2) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength Combined) (PK3)
Number analyzed (Participants) | 23 | 20
hours (h) | 23.342 [20.472 to 26.615] | 22.337 [19.574 to 25.490]

43. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf) as Measured by the Two-stage Chromogenic Assay for PK2 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: AUCinf is area under the concentration-time curve from time zero to infinity.
Time Frame: Pre-dose and post dose at: 0.5 hour (hr), 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK2) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK2)
Number analyzed (Participants) | 11 | 12
IU*h/dL | 2599.2 [2257.2 to 2993.1] | 2951.9 [2376.1 to 3667.2]

44. Secondary Outcome: Incremental Recovery (IR) of rFVIIIFc as Measured by the Two-stage Chromogenic Assay for PK2 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: as for outcome 16
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL per IU/kg
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK2) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK2)
Number analyzed (Participants) | 11 | 12
IU/dL per IU/kg | 3.225 [2.643 to 3.936] | 3.278 [2.835 to 3.792]

45. Secondary Outcome: Maximum Activity (Cmax) of rFVIIIFc as Measured by the Two-stage Chromogenic Assay for PK2 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: Cmax is defined as maximum activity of rFVIIIFc.
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK2) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK2)
Number analyzed (Participants) | 11 | 12
IU/dL | 161.38 [132.29 to 196.88] | 163.97 [141.78 to 189.64]

46. Secondary Outcome: Half-life (t½) of rFVIIIFc as Measured by the Two-stage Chromogenic Assay for PK2 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: Time required for the concentration of the drug to reach half of its original value.
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: Hours (h)
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK2) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK2)
Number analyzed (Participants) | 11 | 12
Hours (h) | 16.687 [14.593 to 19.080] | 19.595 [15.680 to 24.488]

47. Secondary Outcome: Clearance (CL) of rFVIIIFc as Measured by the Two-stage Chromogenic Assay for PK2 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: as for outcome 19
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: mL/h/kg
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK2) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK2)
Number analyzed (Participants) | 11 | 12
mL/h/kg | 1.9236 [1.6705 to 2.2152] | 1.6938 [1.3634 to 2.1043]

48. Secondary Outcome: Volume of Distribution at Steady State (Vss) of rFVIIIFc as Measured by the Two-stage Chromogenic Assay for PK2 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: as for outcome 20
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK2) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK2)
Number analyzed (Participants) | 11 | 12
mL/kg | 41.15 [34.50 to 49.07] | 42.83 [37.33 to 49.15]

49. Secondary Outcome: Mean Residence Time (MRT) of rFVIIIFc as Measured by the Two-stage Chromogenic Assay for PK2 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: as for outcome 21
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: hours (h)
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK2) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK2)
Number analyzed (Participants) | 11 | 12
hours (h) | 21.391 [17.713 to 25.833] | 25.287 [20.729 to 30.847]

50. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf) as Measured by the Two-stage Chromogenic Assay for PK3 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: AUCinf is area under the concentration-time curve from time zero to infinity.
Time Frame: Pre-dose and post dose at: 0.5 hour (hr), 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK3) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK3)
Number analyzed (Participants) | 8 | 12
IU*h/dL | 2646.8 [1891.8 to 3703.0] | 2829.4 [2235.7 to 3580.8]

51. Secondary Outcome: Incremental Recovery (IR) of rFVIIIFc as Measured by the Two-stage Chromogenic Assay for PK3 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: as for outcome 16
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL per IU/kg
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK3) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK3)
Number analyzed (Participants) | 11 | 12
IU/dL per IU/kg | 2.891 [2.413 to 3.464] | 3.016 [2.597 to 3.504]

52. Secondary Outcome: Maximum Activity (Cmax) of rFVIIIFc as Measured by the Two-stage Chromogenic Assay for PK3 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: Cmax is defined as maximum activity of rFVIIIFc.
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: The PKAS is defined as all participants with evaluable PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK3) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK3)
Number analyzed (Participants) | 11 | 12
IU/dL | 144.58 [120.66 to 173.25] | 151.15 [130.34 to 175.28]

53. Secondary Outcome: Half-life (t½) of rFVIIIFc as Measured by the Two-stage Chromogenic Assay for PK3 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: Time required for the concentration of the drug to reach half of its original value.
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Hours (h)
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK3) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK3)
Number analyzed (Participants) | 8 | 12
Hours (h) | 16.945 [13.793 to 20.818] | 17.522 [14.213 to 21.601]

54. Secondary Outcome: Clearance (CL) of rFVIIIFc as Measured by the Two-stage Chromogenic Assay for PK3 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: as for outcome 19
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: milliliter per hour per kilogram(mL/h/kg
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK3) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK3)
Number analyzed (Participants) | 8 | 12
milliliter per hour per kilogram(mL/h/kg | 1.8891 [1.3502 to 2.6429] | 1.7709 [1.3989 to 2.2419]

55. Secondary Outcome: Volume of Distribution at Steady State (Vss) of rFVIIIFc as Measured by the Two-stage Chromogenic Assay for PK3 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: as for outcome 20
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK3) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK3)
Number analyzed (Participants) | 8 | 12
mL/kg | 41.78 [30.70 to 56.87] | 39.82 [35.98 to 44.06]

56. Secondary Outcome: Mean Residence Time (MRT) of rFVIIIFc as Measured by the Two-stage Chromogenic Assay for PK3 at Different Vial Strengths (1000 and 6000 IU/Vial)
Description: as for outcome 21
Time Frame: Pre-dose and post dose at: 0.5 hr, 1 hr, 6 hr, 24 hr, 48 hr, 72 hr and 96 hr
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: hours (h)
Arm/Group | 15K rFVIIIFc (1000 IU/Vial Strength) (PK3) | 15K rFVIIIFc (6000 IU/Vial Strength) (PK3)
Number analyzed (Participants) | 8 | 12
hours (h) | 22.119 [17.717 to 27.614] | 22.483 [18.532 to 27.277]

57. Secondary Outcome: Development of Inhibitors as Measured by the Nijmegen-modified Bethesda Assay
Description: An inhibitor test result greater than or equal to (>=)0.6 Bethesda units [BU]/mL, confirmed on 2 separate samples drawn 2 to 4 weeks apart, was considered positive. The test was performed by the central laboratory using the Nijmegen-modified Bethesda Assay. An exact 95% confidence interval (CI) for the percentage of participants with a confirmed inhibitor was calculated using the Clopper-Pearson method for a binomial proportion. Percentage of participants with confirmed inhibitor development was summarized overall.
Time Frame: At screening and predose on Day 1, 13 and 26 weeks after PK2 injection or at Early Termination (Approximately 43 weeks)
Population: The population analyzed included all participants who received at least 1 dose of rFVIIIFc.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 2K/15K rFVIIIFc (1000/6000 IU/Vial Strength)- All Participants: All participants received rFVIIIFc (1000 IU/vial strength), 50 IU/kg, manufactured in 2K (2000 liter bioreactor scale) for PK1. At PK1, participants were randomized to receive rFVIIIFc (1000 or 6000 IU/vial strength), 50 IU/kg, manufactured in 15K (15000 liter bioreactor scale) for PK2. Following PK2 assessments, participants received prophylactic treatment with any of 5 available 15K vial strengths during the treatment phase. After 13 weeks of treatment with 15K rFVIIIFc, participants were re-evaluated at PK3 at the same vial strength as in PK2. A minimum of 120 hours of washout was observed prior to the PK2 assessment. Following the PK3 assessment, participants were resumed to treatment in the Treatment Period until they complete a total of at least 26 weeks of treatment.
Arm/Group | 2K/15K rFVIIIFc (1000/6000 IU/Vial Strength)- All Participants
Number analyzed (Participants) | 24
percentage of participants | 0 [0 to 14.25]

58. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) at 15K Manufacturing Scale
Description: An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. Number of Participants with TEAEs were summarized overall.
Time Frame: Approximately 43 weeks
Population: The population analyzed included all participants who received at least 1 dose of rFVIIIFc at 15k manufacturing scale.
Measure: Count of Participants; unit: Participants
Groups:
- 15K rFVIIIFc (1000 and 6000 IU/Vial Strength): Participants who received 2K rFVIIIFc 1000 IU/vial (50 IU/kg) for PK1 were randomized to receive rFVIIIFc (1000 or 6000 IU/vial strength), 50 IU/kg, manufactured in 15K (15000 liter bioreactor scale) for PK2. Following PK2 assessments, participants received prophylactic treatment with any of 5 available 15K vial strengths during the treatment phase. After 13 weeks of treatment with 15K rFVIIIFc, participants were re-evaluated at PK3 at the same vial strength as in PK2. A minimum of 120 hours of washout was observed prior to the PK2 assessment. Following the PK3 assessment, participants were resumed to treatment in the Treatment Period until they complete a total of at least 26 weeks of treatment.
Arm/Group | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength)
Number analyzed (Participants) | 23
Participants | 10

59. Secondary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (TESAEs) at 15K Manufacturing Scale
Description: An SAE is any untoward medical occurrence that at any dose: results in death or in the view of the Investigator, places the participant at immediate risk of death (a life-threatening event); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; or results in a congenital anomaly/birth defect. All major surgeries will be reported as SAEs. An SAE may also be any other medically important event that, in the opinion of the Investigator, may jeopardize the participant or may require intervention to prevent one of the other outcomes listed in the SAE definition. Number of participants with TESAEs were summarized overall.
Time Frame: Approximately 43 weeks
Population: The population analyzed included all participants who received at least 1 dose of rFVIIIFc at 15k manufacturing scale.
Measure: Count of Participants; unit: Participants
Arm/Group | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength)
Number analyzed (Participants) | 23
Participants | 0

ADVERSE EVENTS:
Time Frame: Approximately 43 weeks
Description: The Safety Population included all participants who received at least 1 dose of rFVIIIFc. Adverse events are reported based on the overall number of participants treated with 2K rFVIIIFc at 1000 IU/vial strength (PK1 assessment period and Intermediate period) and 15K rFVIIIFc at 1000 and 6000 IU/vial strength (PK2 assessment period and Treatment Period).
Arm/Group | 2K rFVIIIFc (1000 IU/Vial Strength) (PK1) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 0/24 | 3/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2K rFVIIIFc (1000 IU/Vial Strength) (PK1) (N=24) | 15K rFVIIIFc (1000 and 6000 IU/Vial Strength) (N=23)
Headache (Nervous system disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2015-09-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT02502149/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/49/NCT02502149/SAP_001.pdf